CLINICAL TRIAL: NCT02587559
Title: Effectiveness of Manual Therapy and Exercise in the Management of Glenohumeral Osteoarthritis: A Randomized Controlled Trial
Brief Title: Effectiveness of Manual Therapy and Exercise in Shoulder OA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not recruit subjects as they routinely chose surgical option
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 042015-091
Record Dates: First submitted 2015-10-20; First posted 2015-10-27 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis
Keywords: physical therapy
MeSH Terms: conditions — Osteoarthritis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): usual medical advice regarding symptomatic control and activity modification
- Experimental (Experimental): Six visits of physical therapy to provide manual therapy and therapeutic exercise
  Interventions: Procedure: physical therapy

INTERVENTIONS:
Procedure: physical therapy — application of manual therapy techniques to upper extremity along with therapeutic exercise procedures to the axioscapular and rotator cuff musculature
  Arms: Experimental

SUMMARY:
Approximately 60 subjects from a sample of convenience diagnosed with shoulder arthritis will be randomized into a two groups. The control group will receive usual medical advice and the experimental group will be referred to physical therapy for eight visits over 4-week period of time. At one month, two months, and one year the pain, function, and patient satisfaction will be compared between the two groups.

DETAILED DESCRIPTION:
This study will be a pragmatic, prospective, single blind, randomized controlled trial. Stratified randomization will be performed to account for those patients that necessitate a subacromial corticosteroid injection prior to or during the physical therapy intervention. The diagnosis of primary glenohumeral osteoarthritis will be confirmed by the orthopedic surgeon involved in the study. All subjects will have radiographs at the time of initial evaluation (standard medical practice) and magnetic resonance imaging will only be required at the discretion of the orthopedic surgeon when this modality is necessary to rule out other shoulder pathologies of concern.

This study will use a convenient sample of consecutive subjects who meet all inclusion criteria and present to the shoulder service physicians at UT Southwestern outpatient clinic with a primary compliant of shoulder pain and stiffness. If appropriate for the study, the subjects will be referred to physical therapy for additional assessment and care. If interested in participation, each potential subject will be educated regarding the purpose and logistics of the study and asked to enroll via informed consent.

Approximately 25 of the 50 subjects will be seen in the clinic for 6 visits within a 4 week time frame. All subjects will return for follow-up or phone call at 4, 8, and 52 weeks for final data collection and outcomes assessment. The last follow-up assessment at one year will be via phone contact. For those attending physical therapy, the duration of the visits, 1-6, will last from 30-60 min. The final visit, visit 9, will take 15-30 minutes. The phone call on the tenth interaction will last 5-10 minutes.

Session 1: Participant Enrollment - Obtainment of consent, HIPPA and health screen. Baseline dependent variable data will be collection and the subjects will be randomly allocated to one of the treatment groups. One group will receive usual medical advice including tips on posture, activity modifications, and symptom control. The other group will initiate the program of physical therapy outlined below. Subjects allocated to the physical therapy treatment arm will proceed to a standard physical therapy visit in which they will be instructed in the initial exercise training and educated on the use exercise log for assessment of compliance.

Session 2-6 (within 4 weeks after session 1): All patients in the experimental group will receive standardized physical therapy intervention to treat shoulder osteoarthritis including manual therapy (no more than 2 units, <37 minutes) and standard flexibility and range of motion exercises. Patient's will also undergo an in clinic assessment of compliance of their exercise program and appropriate progression of the shoulder strengthening exercises will be provided. Patients in the control group will not participate in sessions 2-5.

Independent Variable:

Group 1 Intervention- manual physical therapy and strengthening exercises to the entire upper quarter, flexibility exercises, range of motion exercises, and usual medical advice.

Manual Therapy: joint mobilization to anterior, posterior, and inferior capsule as indicated at discretion of treating physical therapist

Shoulder Exercise Training:

1. Adducted ER with towel roll in sitting or standing ("no-money" exercise with concurrent external rotation)
2. Supine or standing boxer punch for serratus
3. Short arc military press progressing to flexion or scaption as tolerated
4. Subscapularis isolation via seated narrow grip internal rotation row
5. Horizontal abduction in neutral (wide grip rows)

   * Compliance to the home exercise program will be assessed using a daily log.
   * All therapeutic exercises with include theraband resistance performed 2-3x20/daily

Session 6 (4 weeks after Session 1): Post-Intervention Data Collection and finalization of the exercise training and self-mobilization protocol for the experimental group. The control group will return for a repeat of baseline testing.

Session 7 (8 weeks after Session 1): Post-Intervention Data Collection - Re-assessment of dependent variables.

Session 8 (one year after enrollment): Phone call to collect outcome assessment data

Dependent Variables:

Primary

1. Numerical pain rating scale at baseline day 28, day 56, and day 365 during scapular plane shoulder elevation
2. Functional Outcome Score: American Shoulder and Elbow Surgeon scale (ASES) questionnaire and Simple Shoulder Test (SST)

Secondary

1. Patient's Global Rating of Change (15 point ordinal scale ranging from -7 to +7)
2. Patient self-reported global percentage of improvement (0-100%)
3. Tampa Scale for Kinesiophobia score
4. Pittsburgh Sleep Quality Index score
5. Internal and External Rotation Range of Motion
6. Scapular Elevation strength via manual muscle test

ELIGIBILITY:
Inclusion Criteria:

* over 50 years of age
* Osteoarthritis > Grade 3 on the Kellgren-Lawrence scale
* Presence of at least two of the following findings:
* morning stiffness that resolves within 60 minutes
* pain > 3/10 on a numerical pain rating scale
* asymmetrical mobility in either contralateral elevation and/or glenohumeral rotation, or notable crepitus with active motion.

Exclusion Criteria:

* medical co-morbidities (diabetes and rheumatoid arthritis)
* adhesive capsulitis
* fractures
* scapulothoracic paresis
* surgery in past year
* inability to speak English language

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Functional Level Change | change in function from baseline to two months
  self-report outcome score via American Shoulder Elbow Surgeon's scale and Simple Shoulder Test

SECONDARY OUTCOMES:
Global Rating of Change | change in rating from baseline to two months
  scale of patient satisfaction
Pittsburgh Sleep Quality Index | change in sleep quality from baseline to two months
  sleep quality assessment

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Smith, PhD, Study Chair — University of Texas Southwestern Medical Center; Edward Mulligan, DPT, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States